CLINICAL TRIAL: NCT04600674
Title: Delayed Cord Clamping in Rhesus Disease of the Newborn: A Randomized Clinical Trial
Brief Title: Delayed Cord Clamping in Rhesus Disease of the Newborn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Shaimaa Reda Abdelmaksoud, M.D. (Lecturer), Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC 1-10-2020
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Rhesus Isoimmunization
Keywords: Rhesus Disease; Newborn
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- delayed cord clamping (Experimental): DCC performed at 60 sec after birth
  Interventions: Procedure: Delayed cord clamping
- early cord clamping (Experimental): ECC performed at 15 sec after birth
  Interventions: Procedure: Early cord clamping

INTERVENTIONS:
Procedure: Delayed cord clamping — DCC performed at 60 sec after birth
  Arms: delayed cord clamping
Procedure: Early cord clamping — ECC performed at 15 sec after birth
  Arms: early cord clamping

SUMMARY:
The objective of this clinical trial is to investigate the effects of delayed cord clamping on hyperbilirubinemia, the need for phototherapy, neonatal intensive care (NICU) admission

DETAILED DESCRIPTION:
The study will include term or preterm infants born to Rh negative mother.

The enrolled infants will be randomized into two groups:

Group (1) will include infants with delayed cord clamping performed at 60 sec after birth Group (2) will include infants with early cord clamping within 15 seconds.

History and examination The data on the gender, gestational age, birth weight, length, head circumference, 5- minute Apgar scores, presence of jaundice requiring phototherapy or exchange transfusion, need for admission in neonatal intensive care unit, the presence of respiratory distress (RR > 60 breath per minute) ,and length of hospitalization will be recorded.

The enrolled infants will be followed either with their mothers in the nursery or in NICU. Regarding the mothers; maternal age, maternal weight, any diseases, medication, and mode of delivery, and postpartum hemorrhage requiring blood transfusion will be recorded.

ELIGIBILITY:
Inclusion Criteria:

- term or preterm infants born to Rh negative mother

Exclusion Criteria:

* Infants with Rh negative factor
* major congenital malformation
* fetal hydrops
* short umbilical cord less than 25cm
* nuchal cord
* multiple gestation
* unstable maternal hemodynamic condition
* placenta abruption
* placenta previa
* uterine rupture
* denied to participate
* depressed neonates who will require immediate resuscitation

Max Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Hematocrit value | 2 hours
  Hematocrit will be measured at 2 hours of life (percent %)

SECONDARY OUTCOMES:
Bilirubin level | 24 hours
  Bilirubin level will be measured at 24 hours of life (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Ramadan A Mahmoud, MD, Study Chair — Sohag Faculty of Medicine, Sohag University; Rana A Khashaba, MD, Study Chair — Benha Faculty of Medicine, Benha University; Walid M Tawfik, MD, Study Chair — Benha Faculty of Medicine, Benha University
Locations (1):
- Benha University Hospital, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garabedian C, Rakza T, Drumez E, Poleszczuk M, Ghesquiere L, Wibaut B, Depoortere MH, Vaast P, Storme L, Houfflin-Debarge V. Benefits of Delayed Cord Clamping in Red Blood Cell Alloimmunization. Pediatrics. 2016 Mar;137(3):e20153236. doi: 10.1542/peds.2015-3236. Epub 2016 Feb 18. PMID 26908660
- [Background] Vural I, Ozdemir H, Teker G, Yoldemir T, Bilgen H, Ozek E. Delayed cord clamping in term large-for-gestational age infants: A prospective randomised study. J Paediatr Child Health. 2019 May;55(5):555-560. doi: 10.1111/jpc.14242. Epub 2018 Oct 4. PMID 30288843